CLINICAL TRIAL: NCT04472572
Title: Expanded Access to Convalescent Plasma for the Treatment of Patients With COVID-19
Brief Title: Expanded Access to Convalescent Plasma for Treatment of COVID-19
Status: No longer available | Type: Expanded Access
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: Pro2020-0663
Record Dates: First submitted 2020-07-14; First posted 2020-07-15 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: Coronavirus; Covid19; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Convalescent Plasma — Fresh or frozen plasma will be infused one time to patients with COVID-19 infection

SUMMARY:
This expanded access program will provide access to investigational convalescent plasma for patients at Hackensack University Medical Center infected with SARS-CoV-2 who have severe or life-threatening COVID-19, or who are judged by a healthcare provider to be at high risk of progression to severe or life-threatening disease.

DETAILED DESCRIPTION:
This expanded access program will provide access to investigational convalescent plasma for patients at Hackensack University Medical Center infected with SARS-CoV-2 who have severe or life-threatening COVID-19, or who are judged by a healthcare provider to be at high risk of progression to severe or life-threatening disease. Following enrollment on the protocol and provision of informed consent, patients will be transfused with approximately 200-500 mL of ABO compatible convalescent plasma obtained from individuals who have recovered from documented infection with SARS-CoV-2 and who have been found to have high anti-SARS-CoV2 titers. Safety information collected will include serious adverse events judged to be related to the administration of convalescent plasma. Other information to be collected retrospectively will include patient demographics, resource utilization (total length of stay, days in ICU, days intubated, and survival to discharge from the facility.

ELIGIBILITY:
Inclusion Criteria:

1. Age at least 18 years
2. Laboratory confirmed diagnosis of infection with SARS-CoV-2
3. Admitted to the hospital for the treatment of COVID-19 complications
4. Severe or life threatening COVID-19, or judged by the treating provider to be at high risk of progression to severe or life-threatening disease
5. Informed consent provided by the patient or healthcare proxy
6. Severe COVID-19 is defined by one or more of the following:

   * dyspnea
   * respiratory frequency ≥ 30/min
   * blood oxygen saturation ≤ 93%
   * partial pressure of arterial oxygen to fraction of inspired oxygen ratio < 300
   * lung infiltrates > 50% within 24 to 48 hours

Life-threatening COVID-19 is defined as one or more of the following:

* respiratory failure/mechanical ventilation
* septic shock
* multiple organ dysfunction or failure

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michele Donato, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

REFERENCES:
- [Background] Roback JD, Guarner J. Convalescent Plasma to Treat COVID-19: Possibilities and Challenges. JAMA. 2020 Apr 28;323(16):1561-1562. doi: 10.1001/jama.2020.4940. No abstract available. PMID 32219429
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Ko JH, Seok H, Cho SY, Ha YE, Baek JY, Kim SH, Kim YJ, Park JK, Chung CR, Kang ES, Cho D, Muller MA, Drosten C, Kang CI, Chung DR, Song JH, Peck KR. Challenges of convalescent plasma infusion therapy in Middle East respiratory coronavirus infection: a single centre experience. Antivir Ther. 2018;23(7):617-622. doi: 10.3851/IMP3243. Epub 2018 Jun 20. PMID 29923831
- [Background] https://www.fda.gov/vaccines-blood-biologics/investigational-new-drug-ind-or-device-exemption-ide-process-cber/investigational-covid-19-convalescent-plasma-emergency-inds